CLINICAL TRIAL: NCT02331654
Title: Spinal Direct Current Stimulation Effects on Pain in Multiple Sclerosis: Clinical and Neurophysiological Assessment and Evaluation of Endocannabinoid System Activity
Brief Title: Spinal Direct Current Stimulation Effects on Pain in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2786/13
Record Dates: First submitted 2014-12-16; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Multiple Sclerosis
Keywords: Chronic pain; Direct Current Stimulation
MeSH Terms: conditions — Multiple Sclerosis; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Treatment (Experimental): Anodal DC stimulation (2 mA, 20 min) will be delivered by a constant direct current electrical stimulator connected to a pair of electrodes: the anode will be placed on the thoracic spinal cord (over the spinal process of the tenth thoracic vertebra) and the cathode (reference) above the right shoulder. Stimulating electrodes will be thick (6 mm), rectangular pieces of saline-soaked synthetic sponge. The sDCS polarity (anodal) will refer to the electrode over the spinal cord.
  Interventions: Other: Experimental treatment
- Placebo treatment (Placebo Comparator): For sham sDCS (placebo), electrodes will be placed as for active stimulation, but the stimulator will automatically turn off after 10 s.
  Interventions: Other: Placebo treatment

INTERVENTIONS:
Other: Experimental treatment — Anodal DC stimulation (2 mA, 20 min) will be delivered by a constant direct current electrical stimulator connected to a pair of electrodes
  Arms: Experimental Treatment
Other: Placebo treatment — Electrodes will be placed as for active stimulation, but the stimulator will automatically turn off after 10 s
  Arms: Placebo treatment

SUMMARY:
Pain represents one of the most common symptoms of Multiple Sclerosis (MS) that can seriously affect patient health-related quality of life.

Central neuropathic pain, the main form of pain in MS patients, represents a significant clinical problem, in consideration of its poorly responsiveness to available therapies.

Direct Current Stimulation (tDCS) is a non-invasive, well-tolerated procedure with an high and well documented neuromodulation activity at Central Nervous System (CNS) level. First evidences obtained by animal, neurophysiological and clinical studies suggested its potential efficacy in neuropathic pain treatment.

In particular spinal DCS (sDCS) has been proven to modulate Nociceptive Withdrawal Reflex (NWR), an objective and sensitive tool to explore pain processing at the Spinal Level and recommended by European Federation of Neurological Society (EFNS) to evaluate the analgesic effect of treatments. In this order of view the investigators' objective is to investigate sDCS efficacy in MS neurophatic pain treatment applying validated clinical scales, neurophysiological acquisitions and specific biological marker dosages.

DETAILED DESCRIPTION:
The investigators plan to recruit, at the IRCCS Neurological National Institute C. Mondino, 60 consecutive patients with definite Multiple Sclerosis (MS) according to 2005 McDonald criteria in a follow-up procedure that includes a general and neurological evaluation scored according to the Expanded Disability Status Scale of Kurtzke and its functional systems.

Relapsing-remitting (RR), secondary-progressive (SP) and primary-progressive (PP) MS patients, affecting by neuropathic or nociceptive chronic pain conditions in accord to 1994 International Association for the Study of Pain (IASP)classification, will be recruited. Patients complaining any form of headache will be excluded by the study. The investigators will excluded also patients with cognitive impairment (Minimental State Examination - MMSE- <= 21) and psychiatry diseases, in particular depression (Back Depression Inventory Scale - BDI - >15).

Characteristic and intensity of pain symptoms will be collected respectively with validated Italian version of Neuropathic Pain Symptoms Inventory Scale (NPSI) and Numerical Rating Scale (NRS). Spasticity of lower legs, if present, will be clinical assessed with Ashworth Scale and Neurophysiologically evaluated with H/M ratio and Vibratory Inhibition of H-Reflex.

Health-Related Quality of Life (HRQoL) will be assessed by means of the Medical Outcome 36-item Short Form Health Survey (SF-36) whereas the presence and severity of fatigue will be assessed by means of the Fatigue Severity Scale (FSS).

RR patients will be evaluated in stationary phase of the disease that is at least two months after the last clinical relapse and at least one month after the end of a steroidal treatment.

Patients will be consecutive enrolled in the study and randomly assigned to two group: 1. Sham and 2. Anodal Spinal Direct Current Stimulation Treatment, in a double-blind, placebo controlled study design.

Before enrollment, the study protocol will be explained to each subject, and informed written consent will be obtained.

The investigators will proceed as follow:

1. Time of enrollment - T0 First Day

   * Complete clinical evaluation with administration of MMSE and BDI for exclusion criteria
   * Randomized assignment to Anodal or Sham treatment group
   * Administration of NPSI, SF-36, HRQoL e FSS
   * Evaluation of Somatosensory Evoked Potential by Posterior Tibial and Medial Nerve stimulation to investigate the somatosensory pathway involvement.
   * Clinical and Neurophysiological evaluation of Spasticity (if present): Ashworth Scale and H/M ratio and HReflex Vibratory Inhibition.
   * Collection of blood sample to evaluate activity of Fatty Acid Amide Hydrolase (FAAH) in platelets.

   Second Day
   * First Anodal or Sham Direct Current Stimulation Treatment Session (sDCS)
   * Neurophysiological acquisition of Nociceptive Withdrawal Reflex (NWR) and NWR Temporal Summation (see 'Neurophysiological Acquisition' Session for details) before and after 30 and 60 minutes the first sDCS treatment
2. sDCS Treatment After evaluation at T0 patients will undergo 10 daily sDCS treatment, 5 days a week (see sDCS treatment session for details).
3. Evaluation after 10 days of treatment - T1

   * Administration of NPSI, SF-36, HRQoL e FESS
   * Clinical and Neurophysiological evaluation of Spasticity (if present): Ashworth Scale and H/M ratio and HReflex Vibratory Inhibition.
   * Collection of blood sample to evaluate activity of Fatty Acid Amide Hydrolase (FAAH) in platelets.
   * Neurophysiological acquisition of Nociceptive Withdrawal Reflex (NWR) and NWR Temporal Summation
4. Evaluation after 1 month from the end of treatment - T2

   * Administration of NPSI, SF-36, HRQoL e FESS
   * Clinical and Neurophysiological evaluation of Spasticity (if present): Ashworth Scale and H/M ratio and HReflex Vibratory Inhibition.
   * Collection of blood sample to evaluate activity of Fatty Acid Amide Hydrolase (FAAH) in platelets.
   * Neurophysiological acquisition of Nociceptive Withdrawal Reflex (NWR) and NWR Temporal Summation

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting (RR), secondary-progressive (SP) and primary-progressive (PP) MS patients, affected by neuropathic or nociceptive chronic pain conditions in accordance to 1994 IASP (International Association for the Study of Pain) classification

Exclusion Criteria:

* Any form of headache
* Cognitive impairment (Minimental State Examination <= 21)
* Psychiatry diseases, in particular depression (Back Depression Inventory Scale >15)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-06 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
sDCS efficacy in pain as determined by NPSI and NRS scale | 30 days
  Spinal DCS (sDCS) has been proven to modulate Nociceptive Withdrawal Reflex (NWR), an objective and sensitive tool to explore pain processing at the Spinal Level and recommended by European Federation of Neurological Society (EFNS) to evaluate the analgesic effect of treatments.

SECONDARY OUTCOMES:
Central endocannabinoid level as determined by Activity of Fatty Acid Amide Hydrolase (FAAH) in platelets | 30 days
  The endocannabinoid system is involved in descending central pain control and can be modulated by other neurostimulation techniques as transcutaneous electrical nerve stimulation. The investigators suppose that one of the major effect of sDCS is to modulate supraspinal central pain control through activation of endocannabinoid system inducing the analgesic effect. Alteration of endocannabinoid system activity is also involved in other pathological aspects of Multiple Sclerosis as spasms, spasticity and incontinence and to acute and chronic neurodegeneration (anti-oxidant activity and inhibition of glutamate release and signalling). Activity of Fatty Acid Amide Hydrolase (FAAH) in platelets will be quantify.
Spasticity as determined by Ashworth Scale | 30 days
  As sDCS reduces NWR area and as it may modulate endocannabinoid system, the investigators could suppose other positive effects of this treatment in Multiple Sclerosis patients as reduction of painful spasms and spasticity. The investigators will evaluate the effect of sDCS on spasticity, if present, investigating its effect on validate ad hoc scales (Ashworth scale) and on neurophysiological acquisitions (H reflex).

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Sandrini, MD, Principal Investigator — IRCCS Fondazione Istituto Neurologico Nazionale C. Mondino
Locations (1):
- IRCCS Fondazione Istituto Neurologico Nazionale C. Mondino, Pavia, Pavia, Italy

REFERENCES:
- [Background] Solaro C, Brichetto G, Amato MP, Cocco E, Colombo B, D'Aleo G, Gasperini C, Ghezzi A, Martinelli V, Milanese C, Patti F, Trojano M, Verdun E, Mancardi GL; PaIMS Study Group. The prevalence of pain in multiple sclerosis: a multicenter cross-sectional study. Neurology. 2004 Sep 14;63(5):919-21. doi: 10.1212/01.wnl.0000137047.85868.d6. PMID 15365151
- [Background] O'Connor AB, Schwid SR, Herrmann DN, Markman JD, Dworkin RH. Pain associated with multiple sclerosis: systematic review and proposed classification. Pain. 2008 Jul;137(1):96-111. doi: 10.1016/j.pain.2007.08.024. Epub 2007 Oct 24. PMID 17928147
- [Background] Nitsche MA, Seeber A, Frommann K, Klein CC, Rochford C, Nitsche MS, Fricke K, Liebetanz D, Lang N, Antal A, Paulus W, Tergau F. Modulating parameters of excitability during and after transcranial direct current stimulation of the human motor cortex. J Physiol. 2005 Oct 1;568(Pt 1):291-303. doi: 10.1113/jphysiol.2005.092429. Epub 2005 Jul 7. PMID 16002441
- [Background] Ferrucci R, Mameli F, Guidi I, Mrakic-Sposta S, Vergari M, Marceglia S, Cogiamanian F, Barbieri S, Scarpini E, Priori A. Transcranial direct current stimulation improves recognition memory in Alzheimer disease. Neurology. 2008 Aug 12;71(7):493-8. doi: 10.1212/01.wnl.0000317060.43722.a3. Epub 2008 Jun 4. PMID 18525028
- [Background] Fregni F, Thome-Souza S, Nitsche MA, Freedman SD, Valente KD, Pascual-Leone A. A controlled clinical trial of cathodal DC polarization in patients with refractory epilepsy. Epilepsia. 2006 Feb;47(2):335-42. doi: 10.1111/j.1528-1167.2006.00426.x. PMID 16499758
- [Background] O'Connell NE, Wand BM, Marston L, Spencer S, Desouza LH. Non-invasive brain stimulation techniques for chronic pain. A report of a Cochrane systematic review and meta-analysis. Eur J Phys Rehabil Med. 2011 Jun;47(2):309-26. Epub 2011 Apr 14. PMID 21494222
- [Background] Polman CH, Reingold SC, Edan G, Filippi M, Hartung HP, Kappos L, Lublin FD, Metz LM, McFarland HF, O'Connor PW, Sandberg-Wollheim M, Thompson AJ, Weinshenker BG, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2005 revisions to the "McDonald Criteria". Ann Neurol. 2005 Dec;58(6):840-6. doi: 10.1002/ana.20703. PMID 16283615
- [Background] Cruccu G, Anand P, Attal N, Garcia-Larrea L, Haanpaa M, Jorum E, Serra J, Jensen TS. EFNS guidelines on neuropathic pain assessment. Eur J Neurol. 2004 Mar;11(3):153-62. doi: 10.1111/j.1468-1331.2004.00791.x. PMID 15009162
- [Background] Sandrini G, Serrao M, Rossi P, Romaniello A, Cruccu G, Willer JC. The lower limb flexion reflex in humans. Prog Neurobiol. 2005 Dec;77(6):353-95. doi: 10.1016/j.pneurobio.2005.11.003. Epub 2005 Dec 28. PMID 16386347
- [Derived] Berra E, Bergamaschi R, De Icco R, Dagna C, Perrotta A, Rovaris M, Grasso MG, Anastasio MG, Pinardi G, Martello F, Tamburin S, Sandrini G, Tassorelli C. The Effects of Transcutaneous Spinal Direct Current Stimulation on Neuropathic Pain in Multiple Sclerosis: Clinical and Neurophysiological Assessment. Front Hum Neurosci. 2019 Feb 12;13:31. doi: 10.3389/fnhum.2019.00031. eCollection 2019. PMID 30809137